CLINICAL TRIAL: NCT04036955
Title: Evaluation of an Innovative Information, Training and Social Support Intervention "INFOSADEM" to Principal Caregivers of Dementia Patients Living at Home. Experimental Study
Brief Title: Evaluation of an Innovative Information, Training and Social Support Intervention "INFOSADEM" to Principal Caregivers of Dementia Patients Living at Home
Acronym: INFOSA-DEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Adelaida Zabalegui Yarnoz, Adelaida Zabalegui Yarnoz, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2014/0317
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Dementia
Keywords: dementia; Alzheimer's disease; patient care; home care
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The INFOSA-DEM programme consists of five, 90-minute informational/training sessions delivered consecutively over one week. Morning or afternoon groups are offered depending on the caregiver's availability. Programme content was developed for use in small groups of 6-8 caregivers. Topics covered in the sessions include basic concepts in dementia and specific issues such as nutrition, rest, medication, physical and cognitive changes, management of behavioural symptoms, affective problems in the patient and informal caregiver, verbal and non-verbal communication techniques, caregiver self-care and information on available resources and community services.
  The sessions are conducted using audio-visual material to facilitate understanding of the content and to encourage active participation among caregivers when talking about their experiences.
  Interventions: Other: INFOSA-DEM
- usual care (No Intervention): Caregivers in the Group control received usual care in the centres where the follow-up was carried out. This consisted of annual or quarterly consultations with a health professional (GP, geriatrician or neurologist) and, depending on the health centre, a nurse and social worker.Currently, there is no homogenous protocol for all care centres for the patient with high levels of cognitive impairment and dependency.

INTERVENTIONS:
Other: INFOSA-DEM — Caregivers in the intervention group received the INFOSA-DEM programme, together with usual care provided by the participating centres, while caregivers in the CG received usual care in the centres where the follow-up was carried out.
  Arms: intervention group

SUMMARY:
Background: Dementia is an illness that mostly affects people of advanced age and causes disability and dependency. Although the difficulties, a vast number of older people with dementia at our context, are cared for in their own homes by a family member, usually their spouse/partner, son, daughter or companion, but it is well known that this could be one of the main factors of institutionalization. However, home care is an effective option for the health system. This care may be provided over months or years and can have negative effects on the caregivers' health. This article describes the development and implementation of a structured, psychoeducational intervention addressed to informal caregivers of people with dementia cared for at home.

Methods: A quasi-experimental study with repeated observations at 3 and 6 months post-intervention was performed. Intentional sampling and convenience assignment method was used for intervention and control groups. The intervention was structured developed at the beginning of the study, which consists of a multicomponent training, information and emotional support programme of five, 90-minute sessions over one week. The control group received Usual Care. The project was approved by the ethics committee (HCB/2014/0317) and follows the recommendations of the Declaration of Helsinki. Evidence gathered from our research will be published at national and international level.

Discussion: The results of this intervention will support other studies and contribute scientific evidence on the importance of promoting non-pharmacologic interventions in informal caregivers of people with dementia. At the same time, they can be used as the basis for the implementation of psycho educational interventions in home care and in long-term care institutions responsible for monitoring people with dementia; responding to training and information needs, and providing the social support that the caregivers themselves demand.

DETAILED DESCRIPTION:
1. Eligibility Criteria People with a diagnose of dementia, living at home and having an informal caregiver.

   Inclusion criteria
   * People with a diagnose of dementia
   * People older than 65 years old
   * Living at home and receiving public formal care* from Primary Health Care centers.
   * Having an informal caregiver** identified being capable of understand healthcare professional advices (this will be measured by healthcare professional criteria).
   * Cognitive level having a MMSE score lower of 24 .
   * Informed consent signed. *We considered public formal care, the health care team working on Primary Care (being home care or primary care) (GPs,Registered Nurse, Social Worker).

     * We considered informal caregiver the person (family or not) who takes care of the PwD and lives together or visit him/her at least three times a week.

   Exclusion criteria
   * People lower than 65 years old
   * People with a psychiatric symptom or Korsakov sindrome
   * People without informal caregiver identified
2. Outcome measures

   * preparation for care through the Preparedness for Caregiving Scale (PCS)
   * Perceived Competence Scale for Care
   * Inventory Family needs
   * Zarit Burden Scale
   * Katz Index of Independence in Activities of Daily Living
   * positive and negative aspects of care with the Caregiver Reaction assessment (CRA)
   * Perceived Social Support Questionnaire (Duke-UNK )
   * Quality of Life Scale (EQ-5D)
   * General Health Questionnaire (GHQ-12)
   * Resource Utilization Questionnaire for dementia (RUD)
   * Neuropsychiatric Inventory (NPI) .
   * Quality of Life in Alzheimer's Disease (QoL-AD)
   * Charlson Comorbidity Index (CCI)
   * Mini-Mental State Examination (MMSE)
   * Global Deterioration Scale (GDS)

ELIGIBILITY:
Inclusion Criteria:

* People with a diagnose of dementia
* People older than 65 years old
* Living at home and receiving public formal care* from Primary Health Care centers.
* Having an informal caregiver** identified being capable of understand healthcare professional advices (this will be measured by healthcare professional criteria).
* Cognitive level having a MMSE score lower of 24 .

  * We considered public formal care, the health care team working on Primary Care (being home care or primary care) (GPs, Registered Nurse, Social Worker). **We considered informal caregiver the person (family or not) who takes care of the PwD and lives together or visit him/her at least three times a week.

Exclusion Criteria:

* People lower than 65 years old
* People with a psychiatric symptom or Korsakov sindrome
* People without informal caregiver identified

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Preparedness for Caregiving | 2 years
  Preparedness for Caregiving Scale (PCS; 8 items): Assess readiness for tasks and demands of caregiving role. Domains include providing physical care, providing emotional support, setting up in-home support services and deling with the stress of caregiving. Participants are asked to identified how well prepared they feel on a scale from not all prepared (0) to very well prepared (4). Cronbach's Alpha: 0.88-93
positive and negative aspects of care | 2 years
  . Caregiver Reaction Aspects (CRA; 24 items): consists of 24 items in five subscales: self-esteem (range 7-35), lack of family support (range 5-25), financial problems (range 3-15), disrupted schedule (range 5-25) and health problems (range 4-20).
perceived social support | 2 years
  Perceived Social Support Questionnaire (Duke-UNK; 8 items): Instrument to measure the strength of the person's social support network. Cronbach's Alpha: 0.88.
Level of Quality of life: EQ-5D | 2 years
  Quality of Life Scale (EQ-5D): a measure of self-reported quality of life that is applicable to a wide range of health conditions and treatments. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Cronbach's Alpha: 0.87.
FAMILY NEEDS | 2 years
  Family needs inventory
level of burden | 2 years
  Zarit Burden Scale (ZBS; 22 items): a questionnaire developed to measure subjective burden among caregivers. Cronbach's Alpha: 0.92.
Neuropsychiatric Inventory (NPI) | 2 years
  Assess dementia-related behavioral symptoms. Is composed by 10 sub-domains: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, deshinibition, irritability/liability, and aberrant motor activity. Cronbach's Alpha:0.88
degree of independence in activities of daily living | 2 years
  Katz index of Activity of Daily Living (KATZ; 5 items): to assess an older adult's baseline ability to bathe, dress, use the toilet, transfer, remain continent, and feed her- or himself. It's also used for evaluating changes in response to illness. Cronbach's Alpha: 0.87
Competence for care | 2 years
  The Perceived Competence Scale for Care

OTHER OUTCOMES:
level of cognitive deterioration | 2 years
  Global Deterioration Scale (GDS): provides caregivers an overview of the stages of cognitive function for those suffering from a primary degenerative dementia such as Alzheimer's disease. It is broken down into 7 different stages. Stages 1-3 are the pre-dementia stages. Stages 4-7 are the dementia stages. Beginning in stage 5, an individual can no longer survive without assistance.
Comorbidity | 2 years
  Charlson Comorbidity Index (CCI): Assess multiple comorbidity. To complete the Index, patients are asked whether they have a history of medical problems in 12 areas. Among patients with chronic medical conditions, the Index categories were predictive of 1-year mortality and health care costs. Cronbach's Alpha: 0.96.

IPD SHARING:
Plan to Share IPD: No